CLINICAL TRIAL: NCT02281942
Title: Behavioral Interventions to Target Self-Control in Abstinent Nicotine Dependent Smokers
Brief Title: Behavioral Interventions to Target Self-Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Laura Carim Todd, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21DA035877-01A1 (NIH)
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking | interventions — Yoga; Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga (Experimental): Sequential movements in coordination to the breath cycle followed by seated and supine postures to release muscle tension.
  Interventions: Behavioral: Yoga
- Education (Placebo Comparator): A series of 30-minute recordings focused on different aspects of healthy living (e.g. diet, stress).
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Yoga
  Arms: Yoga
Behavioral: Education
  Arms: Education

SUMMARY:
Low self-control has been associated with a number of unhealthy behaviors with low treatment success. Alternative non-pharmacological approaches have the potential for enhancing self-control. This pilot study will investigate if the practice of yoga and/or health and wellness education improve self-control in the context of nicotine addiction, and will set the stage for larger clinical trials using behavioral interventions to supplement or replace existing treatments and increase the rates of recovery from disorders in which low self-control is a susceptibility factor.

ELIGIBILITY:
Inclusion Criteria:

* should smoke a minimum of 10 cigarettes/day
* be fluent speaking and reading English
* in good physical health
* intend to quit smoking
* capable of abstaining from smoking for 12-14 hours
* should have easy daily access to a computer and/or other internet-enabled device

Exclusion Criteria:

* current alcohol or substance use disorder (except nicotine)
* pregnancy
* history of psychosis or bipolar disorder
* current use of a behavioral or pharmacologic tobacco treatment
* any untreated medical or psychiatric condition that might compromise their safety during participation in the study (e.g. high blood pressure, diabetes, BMI >35)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Time (minutes) to first smoke after 12-hour abstinence | Assessed 1 week after visit 1 during a 2-hour abstinence reinforcement session

CONTACTS AND LOCATIONS:
Overall Officials: Laura Carim Todd, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States